CLINICAL TRIAL: NCT06656793
Title: Impact of Real-Time Ultrasound-Guided Spinal Anesthesia Versus Landmark-Guided Spinal Anesthesia on Anesthesia Procedural Time
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Tianzhu Liu, Principal Investigator, Tongji Hospital
Other Study IDs: Tongji Hospital102114-5
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Spinal Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- RT-SA: Real-Time Ultrasound-Guided Spinal Anesthesia
- LM-SA: Landmark-Guided Spinal Anesthesia

SUMMARY:
Intraspinal anesthesia, traceable to the late 19th century, involves injecting local anesthetics into the spinal canal to block nerve signals, relieving pain and relaxing muscles for surgery. Compared with general anesthesia, it has advantages: smaller impact on the central nervous system, lower drug dosage (reducing systemic poisoning risk), precise block plane control (protecting respiratory/cardiac function), and benefits for mothers and fetuses.

However, traditional blind puncture faces challenges in special patients (obese, post-spinal surgery, or pathological cases). It relies on "loss of sensory resistance," prone to misjudgment, leading to dura rupture or spinal cord injury. Obese pregnant women have hard-to-palpate spinous processes; the elderly have ligament calcification/narrowed intervertebral spaces, affecting positioning and ultrasound imaging.

Ultrasound guidance has advanced since 1984 (first used to measure epidural space depth, reducing complications). It aids obese pregnant women in locating spinal structures, guides pediatric epidural catheter placement, and improves first-attempt success with better resolution. Adjusting the ultrasound probe to a sagittal midline inner oblique angle solves imaging issues in elderly patients.

Clinically, 24G/25G fine needles for ultrasound-guided lumbar puncture may deform; the "needle-in-a-needle" technique (using a larger guide needle) reduces tissue damage and accidental dura puncture, while minimizing skin punctures.

Small-sample studies confirm ultrasound's value in vertebral localization and real-time guidance, but the efficacy of ultrasound vs. surface marking remains controversial due to lack of large-sample data. This article provides evidence-based reference via retrospective analysis of 3,597 cases.

DETAILED DESCRIPTION:
The history of intraspinal anesthesia can be traced back to the late 19th century, when attempts were made to perform anesthesia through the spinal canal. Over time, this technique has been improved and refined, allowing local anesthetic drugs to be injected into the spinal canal, temporarily blocking the transmission of signals from the spinal cord and surrounding nerves. This effectively relieves pain in specific parts of the body, relaxes muscles, and meets the surgical needs. Therefore, intraspinal anesthesia has become an important part of modern anesthesia.

Compared with general anesthesia, intraspinal anesthesia has unique technical advantages: Firstly, it mainly acts on the spinal cord, having a smaller impact on the central nervous system; Secondly, the required drug dosage is smaller, less likely to cause systemic drug poisoning reactions; Moreover, by precisely controlling the block plane, it can maximize the protection of the patient's respiratory function and cardiac autonomic function, while avoiding respiratory system damage or infection, as well as cardiovascular and cerebrovascular complications caused by ventilation control or systemic drug stimulation. Furthermore, since the local anesthetic only acts on the spinal cord during the specific physiological delivery process for the mother, intraspinal anesthesia is very beneficial for both the mother and the fetus, making it almost always superior to other anesthesia methods.

However, for some special patients, such as obese patients, those with a history of spinal surgery, or those with pathological changes, the operation of intraspinal anesthesia poses challenges to the traditional blind puncture. The blind puncture method relies on the principle of "loss of sensory resistance", because for such patients, this perception may be misjudged, and multiple punctures may also lead to the rupture of the dura mater or spinal cord injury. In 1984, anesthesiologists first used ultrasound to measure the depth of the epidural space, providing preoperative guidance for the blind puncture operation, and through this improvement, the complications of blind puncture were significantly reduced. Ultrasound also showed advantages in the diagnosis of neonatal epidural hematoma. Although the resolution of the ultrasound images was low at that time, the range of abnormal dura structures was still clearly visible under ultrasound. Obesity in pregnant women is an important factor for blind puncture into the spinal canal. The increase in subcutaneous fat makes it difficult to palpate the spinous processes. In addition, the deep structures within the spinal canal also increase the uncertainty of blind puncture into the spinal canal. Scanning in the sagittal posterior midline approach helps determine the spinous processes, the number of vertebrae, the width of the intervertebral spaces, and the depth of the epidural space, thereby providing specific information about the intraspinal structures before blind puncture. Moreover, ultrasound can guide the placement of epidural catheters in children and confirm the appropriate height of the catheter. In recent years, more and more studies have pointed out that with the improvement of the resolution of ultrasound equipment, the success rate of the first puncture in ultrasound-guided abdominal puncture has significantly increased compared to the blind puncture group. Ultrasound can visualize part of the intraspinal structure and provide a new option for some complex intraspinal punctures. In addition, due to the reduction in the difficulty of intraspinal puncture operations by ultrasound guidance, more anesthesiologists tend to use this technique. For elderly patients, ligament calcification, narrowed intervertebral spaces, and stiff spinal joints can all affect the positioning of the body before spinal puncture and the quality of ultrasound imaging of intraspinal structures. Moreover, since the spinous processes may obstruct the epidural space, the posterior sagittal approach may not clearly display the posterior part of the dura mater. Although the transverse midline approach also reduces the exposure level of ligaments and the influence of spinous bones on the puncture path, the cross-section of ultrasound scanning still needs to pass through the ligament and spinous space required by the traditional blind method. Therefore, for patients with obvious intervertebral space calcification or narrow spinous space, the ultrasound examination of the epidural space still has problems. Based on this consideration, the angle of the ultrasound scan was improved. It was found that positioning the probe at the inner oblique position on the midline of the sagittal plane could effectively avoid these obstacles, thereby making the ultrasound image of the spinal canal clearer. This further reduced the difficulty of spinal canal puncture guided by ultrasound and improved the puncture efficiency. At the same time, the shape of the puncture needle was also clearer, facilitating real-time ultrasound-guided spinal canal puncture.

Currently, the ultrasound-guided spinal subarachnoid anesthesia (lumbar anesthesia) puncture needles we use are generally 24G or 25G fine needles. For ligament calcification or resistant punctures, the fine needle body is prone to deformation or bending. Therefore, we use a larger injection needle as the guiding needle for lumbar anesthesia, that is, the "needle in a needle" technique. This technique avoids the tissue damage caused by directly using the dural puncture needle as the guiding needle and reduces the risk of accidental spinal dural puncture. At the same time, we can directly use the needle tip at the puncture point in the lumbar anesthesia kit for local anesthesia and continue to place it under the skin as the guiding needle after injecting subcutaneous local anesthetic, to avoid multiple skin punctures. With the assistance of the low-frequency ultrasound probe, the straight advancement of the local anesthesia needle can also help us determine the puncture direction.

Previous small sample studies have confirmed that ultrasound can assist in locating the vertebral segment, judging the depth and visibility of the dura mater, and providing real-time guidance for abdominal puncture or epidural catheter insertion. All of the above application methods have been proven to significantly improve the puncture success rate, shorten the puncture time, and reduce the puncture difficulty. However, the differences in the application effects of surface marking positioning and real-time ultrasound guidance in spinal canal anesthesia still remain controversial. Up to now, there is no large sample study comparing the clinical application effects of ultrasound real-time guidance vs. surface marking lumbar anesthesia techniques for analysis.

This article provides an evidence-based medical reference by retrospectively reporting 3597 cases of the clinical application of ultrasound real-time guidance vs. surface marking lumbar anesthesia techniques in patients.

ELIGIBILITY:
Inclusion Criteria:

* None

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who received the real-time needle in needle technique UG-SA between 1 January 2019 and 29 May 2024.
Sampling Method: Non-Probability Sample
Enrollment: 3597 (Actual)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
Door to skin time (Dts) | From 1 January 2019 to 29 May 2024
  The time from when the patient enters the operating room until the skin incision is made.

SECONDARY OUTCOMES:
Operative duration | From the incision to the completion of the surgery
  The duration of operative procedure
Anaesthetic duration | From the beginning of ultrasound guided spinal anesthesia (UG-SA) to the end of anesthesia
  The duration of anesthesia procedure
PACU duration | The time from entering PACU to exiting PACU
  The duration of PACU stay
Blood loss | During operation
  Blood loss during opeartion
Other complications | During operation
  Complications related to spinal anesthesia
Intraspinal dosage of local anesthetics | During operation
  Local anesthetics administrated intraspinal space
Sedation administration (Yes or No) | During operation
  Bolus administration or pumping administration
Remedial opioids (Yes or No) | During operation
  If the patient complains of pain during surgery, remedial opioids are administered intravenously
Vasoactive drugs administration (Yes or No) | During operation
  Vasoactive drugs administrated to avoid HR and BP decreased by more than 20%
Vertebral level of intraspinal puncture | From 1 January 2019 to 29 May 2024
  Intervertebral segment selected by the anesthesiologist for puncture
Time of ultrasound localization | Before ultrasound guided spinal anesthesia (UG-SA) procedure
  Time of ultrasound assessment and localization
Time of UG-SA | From the beginning to the end of the UG-SA
  The procedure time of UG-SA
Upper level of intraspinal block | 15 minutes after UG-SA
  Presented by segmental innervation of spinal nerves
Heart rate, HR | 10, 20, and 30 minutes after UG-SA
  HR data were recorded at 10, 20 and 30 minutes after spinal anesthesia
Systolic blood pressure, SBP | 10, 20, and 30 minutes after UG-SA
  SBP data were recorded at 10, 20 and 30 minutes after spinal anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China